CLINICAL TRIAL: NCT02254720
Title: A Randomised, Single-blind, Placebo-controlled (Within Dose Groups) Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Intravenous Doses (2.5 μg, 7.5 μg, 25 μg, 50 μg, 100 μg, 200 μg, 350 μg, 500 μg Free Cation) BEA 2180 BR in Healthy Male Volunteers With an Additional Arm by Inhalation in One Dose Group (1600 μg)
Brief Title: Safety, Tolerability and Pharmacokinetics of BEA 2180 BR in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1205.5
Record Dates: First submitted 2014-10-01; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Inhalation

ARMS (3):
- BEA 2180 BR IV (Experimental): Rising doses
  Interventions: Drug: BEA 2180 BR solution for infusion
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BEA 2180 BR inhalation (Experimental)
  Interventions: Drug: BEA 2180 BR solution for inhalation; Device: Respimat®

INTERVENTIONS:
Drug: BEA 2180 BR solution for infusion
  Arms: BEA 2180 BR IV
Drug: Placebo — Intravenous infusion
  Arms: Placebo
Drug: BEA 2180 BR solution for inhalation
  Arms: BEA 2180 BR inhalation
Device: Respimat®
  Arms: BEA 2180 BR inhalation

SUMMARY:
Evaluation of safety, tolerability and pharmacokinetics of single rising intravenous doses of BEA 2180 BR; additional exploration of metabolism following inhalation

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male based upon a complete medical history, including the physical examination, regarding vital signs (BP, PR), 12 lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
2. Age ≥21 and ≤50 years
3. BMI ≥18.5 and <29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure (BP), pulse rate (PR), and ECG measurements) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to enrolment in the study or during the study
10. Participation in another trial with an investigational drug within 2 months prior to randomisation
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (regularly more than 40 g alcohol per day for men)
14. Drug abuse
15. Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
16. Excessive physical activities within 1 week prior to randomisation or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of the study centre

    The following exclusion criteria are specific for this study due to the known class side effect profile of anticholinergic drugs:
19. hypersensitivity to tiotropium and/or related drugs of these classes
20. history of narrow-angle glaucoma
21. history of prostatic hyperplasia
22. history of bladder-neck obstruction

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal findings in physical examination | Up to day 12 after drug administration
Number of participants with clinically significant changes in vital signs | Up to day 12 after drug administration
Number of participants with abnormal findings in 12 - lead ECG (electrocardiogram) | Up to day 12 after drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to day 12 after drug administration
Number of participants with adverse events | Up to day 12 after drug administration
Investigator assessed tolerability on a 4-point scale | Up to day 12 after drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours after drug administration
tmax (time from dosing to maximum measured concentration) | Up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 72 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | Up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 72 hours after drug administration
λz (terminal rate constant in plasma) | Up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 72 hours after drug administration
MRT(mean residence time of the analyte in the body) | Up to 72 hours after drug administration
CL (total clearance of the analyte in plasma) | Up to 72 hours after drug administration
Vz (apparent volume of distribution during the terminal phase λz) | Up to 72 hours after drug administration
Vss (apparent volume of distribution at steady state following intravascular administration) | Up to 72 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | Up to 72 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | Up to 72 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | Up to 72 hours after drug administration